CLINICAL TRIAL: NCT02381717
Title: Comparison of Ultrasound Guided Femoral Nerve Blockade and Standard Parenteral Opioid Pain Management Alone in Patients With Hip Fracture in the Emergency Department
Brief Title: Ultrasound Guided Femoral Nerve Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Beatrice Hoffmann, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000304
Record Dates: First submitted 2015-02-27; First posted 2015-03-06 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hip Fracture
Keywords: ultrasound; bupivacaine; femoral nerve block; pain reduction
MeSH Terms: conditions — Hip Fractures | interventions — Bupivacaine; Analgesia; Morphine; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ultra-sound guided femoral nerve block (Experimental): Patients in this arm will receive a bed-side ultrasound guided femoral nerve block with analgesia 0.5% bupivacaine (2mg/kg)
  Interventions: Other: ultra-sound guide; Drug: bupivacaine
- standard of care- IV morphine (Active Comparator): Patients in this arm will have the femoral nerve block block with no ultrasound for guidance with analgesia (IV morphine)
  Interventions: Drug: morphine

INTERVENTIONS:
Other: ultra-sound guide — Patients randomized to this arm will have the femoral nerve block with the guidance of a bedside ultrasound
  Arms: ultra-sound guided femoral nerve block
Drug: bupivacaine
  Other Names: femoral nerve block femoral nerve block with analgesia 0.5% bupivacaine (2mg/kg)
  Arms: ultra-sound guided femoral nerve block
Drug: morphine
  Other Names: femoral nerve block block with no ultrasound for guidance with analgesia (IV morphine)
  Arms: standard of care- IV morphine

SUMMARY:
The goal of the study is to evaluate whether pain control achieved by Ultrasound Guided Femoral Nerve Blockade (USFNB) is equal in efficacy to standard pain management practice of parenteral injection of opioid pain medication in patients presenting to the emergency department (ED) with hip fracture.

DETAILED DESCRIPTION:
In this proposed protocol the investigators will conduct a prospective, randomized control trial comparing the efficacy of Ultrasound Guided Femoral Nerve Blockade (USFNB) versus the standard of care pain management by parenteral injection of opioid pain medication of patients presenting with hip fracture at the BIDMC ED. We hypothesize that USNFB approach will be non-inferior in achieving pain control (efficacy) and superior in the total dose of opioids (lower amount) as compared to the standard protocol. The enrolled population will be randomized 1:1 using a simple balanced randomization scheme.

Participants will be surveyed six times 6 times on a Visual Analog Scale (VAS)* on their pain intensity reduction over 4 hours.

Physicians performing the block will be surveyed promptly following the procedure regarding difficulty performing the block and its efficacy.

Specific Aim #1: The investigators hypothesize that in patients presenting to the ED with hip fracture, USFNB will demonstrate equal efficacy in pain relief with fewer side effects when compared to conventional parenteral opioid therapy. The investigators evaluate this hypothesis by monitoring Visual Analogue Scales (VAS) in patients receiving either USGFNB or opioid therapy over the first 4 hours of observation. The side effects will be noted during the same interval of time.

Specific Aim #2: The investigators hypothesize that in patients presenting to the ED with hip fracture, USFNB will reduce the amount of narcotic used to control pain. The investigators will evaluate this by studying narcotic use over the first 4 hours of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age presenting to the ED with radiographically established intra-, extracapsular hip fracture, able to consent and participate in the study and who have moderate to severe pain (numerical pain score >= 31) at the time of enrollment.

Exclusion Criteria:

* Patients with a previous history of hypersensitivity to local anesthetics,
* Patients who have signs of a local infection at the site of planned needle placement.
* INR > 1.4NOAC use within 48 hours
* Prophylactic Low-Molecular Weight Heparin (LMWH) within 12 hours
* Therapeutic LMWH within 24 hours
* Prophylactic Unfractionated Heparin (5000 Units BID or TID) within 6 hours

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2025-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
pain intensity reduction | 4 hours after initiation of study proceduure
  Evaluation of pain severity and relief will be assessed utilizing a Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Hoffmann, MD PhD, Principal Investigator — Beth Israel Deaconess Medical
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Vincent's Hospital, Worcester, Massachusetts

REFERENCES:
- [Background] Morrison RS, Magaziner J, Gilbert M, Koval KJ, McLaughlin MA, Orosz G, Strauss E, Siu AL. Relationship between pain and opioid analgesics on the development of delirium following hip fracture. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):76-81. doi: 10.1093/gerona/58.1.m76. PMID 12560416
- [Background] Christos SC, Chiampas G, Offman R, Rifenburg R. Ultrasound-guided three-in-one nerve block for femur fractures. West J Emerg Med. 2010 Sep;11(4):310-3. PMID 21079698
- [Background] Baker BC, Buckenmaier C, Narine N, Compeggie ME, Brand GJ, Mongan PD. Battlefield anesthesia: advances in patient care and pain management. Anesthesiol Clin. 2007 Mar;25(1):131-45, x. doi: 10.1016/j.anclin.2006.12.003. PMID 17400161
- [Background] Fletcher AK, Rigby AS, Heyes FL. Three-in-one femoral nerve block as analgesia for fractured neck of femur in the emergency department: a randomized, controlled trial. Ann Emerg Med. 2003 Feb;41(2):227-33. doi: 10.1067/mem.2003.51. PMID 12548273
- [Background] Malchow RJ, Black IH. The evolution of pain management in the critically ill trauma patient: Emerging concepts from the global war on terrorism. Crit Care Med. 2008 Jul;36(7 Suppl):S346-57. doi: 10.1097/CCM.0b013e31817e2fc9. PMID 18594262
- [Background] Grabinsky A, Sharar SR. Regional anesthesia for acute traumatic injuries in the emergency room. Expert Rev Neurother. 2009 Nov;9(11):1677-90. doi: 10.1586/ern.09.110. PMID 19903026
- [Background] O'Donnell BD, Mannion S. Ultrasound-guided femoral nerve block, the safest way to proceed? Reg Anesth Pain Med. 2006 Jul-Aug;31(4):387-8. doi: 10.1016/j.rapm.2006.04.007. No abstract available. PMID 16857561
- [Background] Marhofer P, Schrogendorfer K, Koinig H, Kapral S, Weinstabl C, Mayer N. Ultrasonographic guidance improves sensory block and onset time of three-in-one blocks. Anesth Analg. 1997 Oct;85(4):854-7. doi: 10.1097/00000539-199710000-00026. PMID 9322469
- [Background] Todd KH. Clinical versus statistical significance in the assessment of pain relief. Ann Emerg Med. 1996 Apr;27(4):439-41. doi: 10.1016/s0196-0644(96)70226-3. No abstract available. PMID 8604855
- [Background] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Background] Platts-Mills TF, Esserman DA, Brown DL, Bortsov AV, Sloane PD, McLean SA. Older US emergency department patients are less likely to receive pain medication than younger patients: results from a national survey. Ann Emerg Med. 2012 Aug;60(2):199-206. doi: 10.1016/j.annemergmed.2011.09.014. Epub 2011 Oct 26. PMID 22032803
- [Background] Bijur PE, Kenny MK, Gallagher EJ. Intravenous morphine at 0.1 mg/kg is not effective for controlling severe acute pain in the majority of patients. Ann Emerg Med. 2005 Oct;46(4):362-7. doi: 10.1016/j.annemergmed.2005.03.010. PMID 16187470
- [Background] Fredrickson MJ, Kilfoyle DH. Neurological complication analysis of 1000 ultrasound guided peripheral nerve blocks for elective orthopaedic surgery: a prospective study. Anaesthesia. 2009 Aug;64(8):836-44. doi: 10.1111/j.1365-2044.2009.05938.x. PMID 19604186
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043